CLINICAL TRIAL: NCT03919305
Title: Cerebral Venous Thrombosis Cohort Study in China Mainland
Acronym: CCC
Status: Not yet recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Other Study IDs: CVT-China
Record Dates: First submitted 2019-04-03; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Cerebral Venous Sinus Thrombosis; Deep Cerebral Vein Thrombosis; Cortical Vein Thrombosis
Keywords: Cerebral venous sinus thrombosis; Deep cerebral vein thrombosis; Cortical vein thrombosis; Cohort study; Real world evidence; Observational study; China mainland; Cerebral venous system thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA detection will be conducted in a ramdom selection of 300 blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was aimed to reveal the clinical features,natural history of the diseases and current therapeutic situations of cerebral venous thrombosis (CVT) in China mainland. Blood samples and cerebrospinal fluid samples will be collected after recruitment to reveal the pathological mechanisms of CVT and identify the biomarkers for CVT.

DETAILED DESCRIPTION:
cerebral venous thrombosis (CVT) is caused by a clot in the cerebral vein, which resulted in an obstruction of the blood outflow. CVT mainly includes cerebral venous sinus thrombosis, deep cerebral vein thrombosis and cortical vein thrombosis. However, the epidemiological features of CVT in China mainland remained obscure. This study was aimed to establish a multicenter cohort recruiting patients with CVT across 31 provinces and municipalities in China mainland. Clinical features,natural history of the diseases and current therapeutic situations will be analyzed to reveal the epidemiological features of CVT. Blood samples and cerebrospinal fluid samples will be collected after recruitment to reveal the pathological mechanisms of CVT and identify the biomarkers for CVT. Patients will be followed-up at 1, 3, 6, 12 months from baseline to evaluate the clinical prognosis and therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

• Cerebral venous sinus thrombosis, deep cerebral vein thrombosis and cortical vein thrombosis diagnosed by digital subtraction angiography (DSA), magnetic resonance venography (MRV), computed tomography venography (CTV) or high-resolution magnetic resonance imaging (HR-MRI).

Exclusion Criteria:

• None of the patient, trustee or immediate family members signed the informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cerebral venous sinus thrombosis, deep cerebral vein thrombosis and cortical vein thrombosis.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Death rate | 1 year from baseline
  A combination of death form of all causes
Functional independence | 1 year from baseline
  Defined as modified Rankin score (0-5) equal to or lower than 2
Recurrence of cerebral venous sinus thrombosis, deep cerebral venous thrombosis and cortical vein thrombosis | 1 year from baseline
  Diagnosed by DSA, MRV, CTV or HR-MRI
Incidence of hemorrhagic complication | 1 year from baseline
  Extracranial hemorrhage (fall in hemoglobin of 2 gram/dl or more within 48 hours) or intracranial hemorrhage
Incidence of sinus wall rupture | 1 year from baseline
Incidence of acute ischemic stroke | 1 year from baseline
Incidence of acute myocardial infarction | 1 year from baseline
Incidence of pulmonary embolism | 1 year from baseline
Incidence of deep venous thrombosis | 1 year from baseline

SECONDARY OUTCOMES:
Incidence of epilepsy | 1 year from baseline
Incidence of allergic reaction | 1 year from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD, PhD, Principal Investigator — Xuanwu Hospital, Beijing

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT03919305/SAP_000.pdf
  • Informed Consent Form (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT03919305/ICF_001.pdf